CLINICAL TRIAL: NCT04098328
Title: Early Feasibility EXperience of Posterior Leaflet RestOration to REduce Mitral Regurgitation (EXPLORE MR)
Brief Title: Early Feasibility EXperience of Posterior Leaflet RestOration to REduce Mitral Regurgitation
Acronym: EXPLORE MR
Status: Terminated | Type: Observational
Why Stopped: Study device refinement
Sponsor: Polares Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 201901
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2022-02

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early feasibility study, single-arm registry design

DETAILED DESCRIPTION:
First-In-Human

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Greater than moderate degenerative or functional mitral regurgitation (Grade 3+ or higher) as confirmed by transesophageal echocardiography (TEE) within 90 days prior to study procedure
3. Patient must present with an STS Score less than 10%
4. High surgical risk for conventional mitral repair or replacement due to morphological criteria (e.g. leaflet or annulus calcifications) as assessed by the local heart team comprised of a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in treating mitral valve disease and heart failure
5. Mitral valve anatomy deemed unsuitable to be treated with an approved edge-to-edge repair system (e.g., retracted posterior leaflet, lack of leaflet tissue, calcified or cleft posterior leaflet) as assessed by the local heart team comprised of a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in treating mitral valve disease and heart failure
6. Patient is approved by an independent Patient Eligibility Committee
7. New York Heart Association (NYHA) Functional Class III or IV
8. Patient willing to participate in study and provide signed EC-approved informed consent.
9. Treating physician and patient agree that patient is able to return for all required post- procedure follow-up visits
10. Women of child-bearing potential have a negative pregnancy test

Exclusion Criteria:

1. Severe tricuspid regurgitation
2. Severe aortic stenosis or insufficiency
3. Severe mitral annulus calcification
4. Diseased mitral anterior leaflet such as flail / prolapse/ heavy calcification
5. Implanted vena cava filter
6. Femoral veins with severe angulation and calcification
7. Contraindication for transesophageal echocardiography (TEE) or MDCT scan.
8. Active infection or endocarditis
9. Previous mitral valve surgery
10. Prior orthotopic heart transplantation
11. Pulmonary artery systolic hypertension > 70mmHg
12. Evidence of intra-cardiac, inferior vena cava (IVC) or femoral venous thrombus
13. Left ventricular ejection fraction (LVEF) < 30%
14. Implant or revision of any pacing device < 30 days prior to intervention
15. Symptomatic coronary artery disease treated < 30 days prior to study procedure
16. Myocardial infarction requiring intervention < 30 days prior to study procedure
17. Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis), hypertrophic or restrictive cardiomyopathies, and constrictive pericarditis
18. Active peptic ulcer or upper gastrointestinal bleeding < 90 days prior to study procedure
19. Stroke < 180 days prior to study procedure
20. Severe renal insufficiency (creatinine > 3.0 mg/dL) or patient requiring dialysis
21. Cardiogenic shock at time of enrolment
22. Hemodynamic instability requiring inotropic support or mechanical heart assistance
23. Concurrent medical condition with a life expectancy of less than 2 years
24. Pregnancy at time of enrolment
25. History of bleeding diathesis or coagulopathy or leukopenia (WBC < 3,000 mcL) or acute anemia (Hb < 9 g/dL) or thrombocytopenia (platelets < 50,000 cells mcL)
26. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel, nitinol, tantalum or allergy to contrast agents that cannot be pre-medicated
27. Severe dementia or lack of capacity due to conditions that result in either inability to provide informed consent for the trial/procedure, prevent independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up assessments
28. Emergency situations
29. Company employees or their immediate family members
30. Patient is under guardianship
31. Patient is participating in another clinical study for which follow-up is currently ongoing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inoperable or high surgical risk patients with symptomatic degenerative or functional mitral regurgitation (Grade 3+ or higher) with mitral valve anatomy deemed unsuitable, or off-label, to be treated with an approved edge-to-edge repair system.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint | 30 days
  All-cause mortality
Improvement from baseline mitral regurgitation | 30 days
  Grade 2+ or less as evaluated by 2D transthoracic echocardiography

SECONDARY OUTCOMES:
Technical success according to MVARC2 criteria | 24 hours
  * Absence of procedure mortality
  * Successful access, delivery and retrieval of investigation delivery system
  * Successful deployment and correct positioning of intended implant(s)
  * Freedom from emergency surgery/re-intervention related to device or access procedure
Procedure success according to MVARC2 criteria | 30 days
  * Absence of procedure mortality or stroke
  * Proper placement and positioning of device
  * Freedom from unplanned re-intervention related to device or access procedure
  * Continued intended safety and performance of the device:
    * No evidence of structural or functional failure
    * No device technical failure issues/complications
    * MR reduction to moderate or less without stenosis
  * Absence of major device or procedure-related SAE:
    * Death
    * Stroke
    * Life-threatening bleed
    * Major vascular complication
    * Major cardiac structural complication
    * No device technical failure issues/complications
    * Stage 2 or 3 AKI
    * MI or coronary ischemia requiring PCI or CABG
    * Shock, heart or respiratory failure requiring IV vasopressors, mechanical intervention or prolonged intubation
    * Valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
Device success according to MVARC2 criteria | 30 days, 6 and 12 months, and 2 - 5 years post treatment
  * Absence of procedure mortality or stroke
  * Proper placement and positioning of device
  * Freedom from unplanned re-intervention related to device or access procedure
  * Continued intended safety and performance of the device:
    * No evidence of structural or functional failure
    * No device technical failure issues/complications
    * MR reduction to moderate or less without stenosis
Patient success according to MVARC2 criteria | 30 days, 6 and 12 months, and 2 - 5 years post treatment
  * Device success
  * Patient returned to pre-procedure setting
  * No rehospitalization or reintervention for mitral regurgitation or heart failure
  * Functional improvement from baseline by one or more NYHA class
  * 6MWT improvement from baseline by 50 metres or more
Rate (%) of major adverse events as defined by MVARC2 criteria | Procedure, discharge/7 days, 30 days, 6 and 12 months, and 2 - 5 years post treatment
  All-cause mortality, hospitalization due to cardiac conditions, stroke or TIA, myocardial infarction, access site and vascular complications, bleeding complications, acute kidney injury up to 7 days post-procedure, and arrhythmias and conduction system disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Brenton, Study Director — Polares Medical; Ulrich Schaefer, MD, Principal Investigator — MarienKrankenhaus & Asklepios Klinik St. Georg, Hamburg (DE); Stephan Windecker, MD, Principal Investigator — Inselspital Bern, Bern (CH)
Locations (3):
- St. Johannes Hospital, Dortmund, Germany
- Switzerland (2):
  - Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne